CLINICAL TRIAL: NCT06527170
Title: Improved Erectile Function After Bariatric Surgery: Role of Testosterone and Other Factors
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Michał Pędziwiatr, Professor, Jagiellonian University
Other Study IDs: JagiellonianU-10
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Bariatric Surgery; Erectile Dysfunction
Keywords: bariatric surgery; erectile dysfunction; obesity
MeSH Terms: conditions — Erectile Dysfunction; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male patients: Male patients undergoing bariatric surgery
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Each patient undergoes bariatric surgery. Each patient is diagnosed before surgery for erectile dysfunction. Similar tests are done 1 year after

SUMMARY:
The prevalence of obesity has risen dramatically worldwide. Beyond its metabolic implications, obesity profoundly impacts sexual health, particularly in males, with erectile dysfunction emerging as a prevalent and distressing comorbidity. Studies show that bariatric surgery alleviates erectile dysfunction. Patients suffering from obesity have lower testosterone levels, which increase after weight-loss surgery. This study aims to investigate the relationship between erectile dysfunction improvement, weight loss and hormonal changes after surgery.

DETAILED DESCRIPTION:
In recent decades, the prevalence of obesity has risen dramatically worldwide, presenting significant public health concerns. Beyond its metabolic implications, obesity profoundly impacts sexual health, particularly in males, with erectile dysfunction (ED) emerging as a prevalent and distressing comorbidity. Obesity exacerbates the risk of ED through complex interplays of physiological and psychological mechanisms. Physiologically, excess adiposity leads to chronic inflammation, endothelial dysfunction, and hormonal imbalances, all of which contribute to impaired vascular health and reduced testosterone levels, key factors in erectile function. Psychologically, body image dissatisfaction and decreased self-esteem associated with obesity can exacerbate sexual performance anxiety and further contribute to ED. Bariatric surgery is an established treatment method for long-term weight loss which also alleviates symptoms of diabetes, hypertension, and other weight-related comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopic sleeve gastrectomy who were qualified according to Guidelines of the International Federation for the Surgery of Obesity and Metabolic Disorders

Exclusion Criteria:

* lack of data during follow-up visit (at 1-year).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients undergoing weight loss surgery at high volume bariatric centre. Male patiens who are sexually active
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
The International Index of Erectile Function score | immediately before surgery and one year after
  6 questions from IIEF official questionnare. Each question is score 1-5.
  Erectile dysfunction (ED) assessed using a validated tool Patient who scored <25 points were considered for further analysis. Each patient was categorized into severity: 25-30 no ED, 19-24 mild ED, 13-18 mild to moderate ED, 7-12 moderate ED, 0-6 severe ED.
  After follow-up, patients with prior ED (<25 IIEF) were assigned to three groups: 1 - no improvement, 2 - symptom alleviation (change in severity category), 3 - ED remission

SECONDARY OUTCOMES:
Weight loss results | one year after surgery
  weight loss (WL) in kg
percentage of excess weight loss (%EWL) | one year after surgery
  Weight loss results
percentage of total weight loss (%TWL) | one year after surgery
  Weight loss results
Testoreone (nmol/l) | immediately before surgery and one year after
  Laboratory test using blood samples
Sex hormone binding (nmol/l) | immediately before surgery and one year after
  Laboratory test using blood samples
Estradiol (pmol/l) | immediately before surgery and one year after
  Laboratory test using blood samples
luteinizing hormone (mIU/ml) | immediately before surgery and one year after
  Laboratory test using blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Michał Pędziwiatr, Prof., Study Director — Jagiellonian University
Locations (1):
- 2nd Department of General Surgery, Jagiellonian University Medical College, Krakow, Małopolska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Malczak P, Wysocki M, Pisarska-Adamczyk M, Strojek J, Rodak H, Lastovetskyi I, Pedziwiatr M, Major P. Influence of Bariatric Surgery on Erectile Dysfunction-a Systematic Review and Meta-Analysis. Obes Surg. 2023 Jun;33(6):1652-1658. doi: 10.1007/s11695-023-06572-9. Epub 2023 Apr 22. PMID 37086370
- [Background] Arolfo S, Scozzari G, Di Benedetto G, Vergine V, Morino M. Surgically induced weight loss effects on sexual quality of life of obese men: a prospective evaluation. Surg Endosc. 2020 Dec;34(12):5558-5565. doi: 10.1007/s00464-019-07356-y. Epub 2020 Jan 14. PMID 31938930
- [Result] Cheng JY, Ng EM. Body mass index, physical activity and erectile dysfunction: an U-shaped relationship from population-based study. Int J Obes (Lond). 2007 Oct;31(10):1571-8. doi: 10.1038/sj.ijo.0803639. Epub 2007 Apr 24. PMID 17452989